CLINICAL TRIAL: NCT00847847
Title: Neuromuscular Transmission in Amyotrophic Lateral Sclerosis
Acronym: NETALS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Association pour la Recherche sur la Sclérose Latérale Amyotrophique (Unknown); Association Française contre les Myopathies (AFM), Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: P080404
Record Dates: First submitted 2009-02-11; First posted 2009-02-19 (Estimated); Last update posted 2012-11-19 (Estimated); Status verified 2009-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: ALS; Motor neuron; Pathophysiology; Neuromuscular junction; Neuromuscular transmission; Microelectrodes
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Other): control subjects with muscle biopsy
  Interventions: Procedure: Anconeus Muscle biopsy
- 1 (Other): ALS patients with muscle biopsy
  Interventions: Procedure: Anconeus Muscle biopsy

INTERVENTIONS:
Procedure: Anconeus Muscle biopsy — Anconeus muscle specimens will be surgically removed. The biopsy will be performed under regional anaesthesia and will require an about 5 cm incision of the skin and muscle fascia from the lateral condyle to over the ridge of the proximal ulna, 3 or 4 cm distal to the tip of the olecranon. A triangular muscle flap will be removed, and then the fascia and skin will be closed with running dissolving suture.

SUMMARY:
Consistent data suggest that neuromuscular transmission is impaired in ALS patients. Neuromuscular junctions dysfunction may appear very early in the disease, as shown by data in animal models. The pathogenesis of this neuromuscular transmission impairment is unknown. Nogo A isoform, a possible marker of the disease over-expressed in skeletal muscle of ALS patients, can be involved. We will characterize the pathophysiological mechanisms implicated using a complete study of the structure and function of the NMJ on muscle biopsies, in a group of 20 ALS patients compared to 10 controls.

DETAILED DESCRIPTION:
Amyotrophic Lateral Sclerosis (ALS) is a progressive neurodegenerative disorder involving motor neurons of the motor cortex, brain stem and spinal cord. Its pathogenesis remains unknown, and the only drug currently available, riluzole, only modestly prolongs survival. Consistent data show that neuromuscular transmission is impaired in patients with ALS. The significance of these abnormalities remains unknown, but recent data suggest that they potentially play a key role in the pathogenesis of the disease. Neuromuscular junctions (NMJs) dysfunction may appear very early in the disease, as shown by data in animal models. The mechanisms of this neuromuscular transmission impairment are unknown. Nogo A belonging to the family of neurite outgrowth inhibitor proteins which is abnormally expressed in skeletal muscle of ALS patients, is probably involved as it has been shown that over-expression of Nogo A in wild-type muscle leads to destabilization of NMJs. A detailed study of the structure and function of the NMJ in ALS patient is mandatory to better characterize the pathophysiological mechanisms implicated.

The aim of this study is to characterize the neuromuscular transmission dysfunction in ALS. For this purpose, we will study the structural and functional features of NMJs on muscle biopsies in a group of 20 ALS patients compared to 10 controls. Using biopsies of a vestigial muscle, the anconeus, we will perform a morphological study of the NMJ, including routine histochemistry, immunohistochemical studies for NMJ major proteins and immune IgG complexes and electron microscopy study. The number of acetylcholine receptors per endplate will be determined by radiolabeled alpha-bungarotoxin binding. Expression levels of Nogo-A will be determined in muscle specimens by western blot. Synaptic transmission at individual NMJs will also be studied ex vivo. We will record membrane potential over time using different nerve stimulation frequencies and we will analyze the properties of the miniature endplate potentials (spontaneous release of acetylcholine) and endplate potentials after stimulation of the nerve (evoked release of acetylcholine). The results of this structural and functional study of NMJ on muscle biopsy will be correlated with surface-EMG and clinical data.

This study will help identifying new mechanisms involved in the pathophysiology of ALS and potential new targets for future treatments.

ELIGIBILITY:
1. ALS patients:

   Inclusion criteria :
   * Aged 18 to 75 (inclusive)
   * Possible, probable (clinically or laboratory) or definite ALS according to the revised El Escorial criteria
   * Duration of the disease of less then 12 months
   * Willing and able to provide a written informed consent
   * With french social insurance affiliation

   Exclusion criteria :
   * Cognitive changes or psychiatric condition, inability to give informed consent
   * patient unable to contact or to be contacted by the investigator in case of emergency
   * women who are pregnant or nursing
   * concomitant medication contraindicating muscular biopsy (platelet suppressive agents if treatment can not medically be stopped 2 weeks before surgical procedure, oral anticoagulant therapy)
   * medical condition contraindicating muscular biopsy (hypo-coagulative disease, allergy to anaesthetic drugs)
   * medical condition susceptible to influence on EMG examination (concomitant neurological or rheumatological disease)
2. Controls:

   * adult patients (minimum 18y) without neuromuscular disease
   * undergoing elbow surgery for local joint or bone disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-03; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Characterization of the neuromuscular transmission dysfunction in ALS by studying the structural and functional features of NMJs on muscle biopsies | within the 15 days after inclusion (month 0 = M0)

SECONDARY OUTCOMES:
Search for correlations between the results of the structural and functional study of neuromuscular junctions on muscle biopsy and surface-EMG and clinical data | at M0, M3, M6

CONTACTS AND LOCATIONS:
Overall Officials: Gaelle Bruneteau, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Bruneteau Gaelle, Paris, France